CLINICAL TRIAL: NCT02459717
Title: Double Blind, Placebo-controlled Trial of a Fermented Milk Containing Multiple Probiotics Strains and Prebiotic Fiber for Constipation Associated With Parkinson's Disease
Brief Title: Pre-biotics and Probiotics for Constipation in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emanuele Cereda (Other)
Collaborators: Fondazione Mondino (Other); Istituti Clinici di Perfezionamento di Milano (Other)
Responsible Party: Sponsor-Investigator, Emanuele Cereda, Co-project Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Organization: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 66/INT/2015
Record Dates: First submitted 2015-05-26; First posted 2015-06-02 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2015-10

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Probiotics; Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics and prebiotic (Experimental): fermented milk (125 grams), containing multiple probiotics strains and prebiotic fiber
  Interventions: Other: Probiotics and prebiotic
- Placebo (Placebo Comparator): pasteurized fermented milk (125 grams) without prebiotics
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probiotics and prebiotic — Patients will receive daily (at breakfast) a fermented milk (125 grams), containing multiple probiotics strains and prebiotic fiber
  Arms: Probiotics and prebiotic
Other: Placebo — Patients will receive daily (at breakfast) a placebo (pasteurized fermented milk without prebiotics)
  Arms: Placebo

SUMMARY:
Constipation is the most frequent (prevalence, about 60%) dysautonomic non motor symptom affecting Parkinson's disease (PD) patients. Unfortunately, limited treatment options have been investigated and are now available for the management of constipation in PD. Preliminary data have suggested that probiotics could be help improving bowel habits but high-quality randomized trials are required in this area. Therefore, the investigators designed a randomized trial to evaluate whether the use of a fermented milk containing multiple probiotics strains and prebiotic fiber have a beneficial effect on constipation in PD compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of constipation according to Roma III criteria
* complete bowel movements per week <3
* total bowel movements per week <6
* written informed consent

Exclusion Criteria:

* report of loose (mushy) or watery stool in the absence of laxative use
* ongoing artificial nutrition
* lactose intolerance
* chronic inflammatory bowel disease
* previous abdominal surgery
* use of anti-cholinergics
* use of antibiotics in the 6 weeks before baseline visit
* Radio- chemotherapy
* Cognitive decline (Mini Mental State Examination <27)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Complete bowel movements | 4 weeks
  Change in the mean number of complete spontaneous bowel movements

SECONDARY OUTCOMES:
Number of bowel movements | 4 weeks
  Change in the mean number of spontaneous bowel movements
Stool consistency | 4 weeks
  Change in mean stool consistency (scored with the use of the 7-point Bristol Stool Form Scale)
Laxative use | 4 weeks
  Change in the mean use of laxative
Treatment satisfaction | 4 weeks
  Satisfaction with the trial medication's ability to relieve constipation symptoms as assessed by a self-rating scale
Treatment continuation | 4 weeks
  Likelihood that patients would continue taking the trial treatment as assessed by a self-rating scale
Increase in one or more complete bowel movements | 4 weeks
  Percentage of patients reporting an increase in one or more complete bowel movements
Frequency of three or more complete bowel movements | 4 weeks
  Percentage of patients reporting three or more complete bowel movements

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Pacchetti, MD, Principal Investigator — IRCCS Istituto Neurologico Mondino
Locations (1):
- IRCCS Istituto Neurologico Mondino, Pavia, Italy

REFERENCES:
- [Derived] Todd CL, Johnson EE, Stewart F, Wallace SA, Bryant A, Woodward S, Norton C. Conservative, physical and surgical interventions for managing faecal incontinence and constipation in adults with central neurological diseases. Cochrane Database Syst Rev. 2024 Oct 29;10(10):CD002115. doi: 10.1002/14651858.CD002115.pub6. PMID 39470206
- [Derived] Barichella M, Pacchetti C, Bolliri C, Cassani E, Iorio L, Pusani C, Pinelli G, Privitera G, Cesari I, Faierman SA, Caccialanza R, Pezzoli G, Cereda E. Probiotics and prebiotic fiber for constipation associated with Parkinson disease: An RCT. Neurology. 2016 Sep 20;87(12):1274-80. doi: 10.1212/WNL.0000000000003127. Epub 2016 Aug 19. PMID 27543643